CLINICAL TRIAL: NCT00250315
Title: Cardiac Dysfunction in Cirrhosis: Cirrhotic Cardiomyopathy Evaluated by Dobutamin MRI.
Brief Title: DOCICAR: Cardiac Dysfunction in Cirrhosis
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Other Study IDs: (KF) 01 270675
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Cirrhosis; Cirrhotic Cardiomyopathy
MeSH Terms: conditions — Fibrosis | interventions — Dobutamine

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Dobutamine

SUMMARY:
Patients with cirrhosis have a altered cardiac response to stress. This study evaluate the cardiac response by MRI during dobutamine stress. Hypothesis: impared increase in cardiac output, cardiac index, ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Non alkoholic cirrhosis

Exclusion Criteria:

* Coma hepaticum
* Primary cardiac diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-11; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Møller, DrMsci, MD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Dahl EK, Moller S, Kjaer A, Petersen CL, Bendtsen F, Krag A. Diastolic and autonomic dysfunction in early cirrhosis: a dobutamine stress study. Scand J Gastroenterol. 2014 Mar;49(3):362-72. doi: 10.3109/00365521.2013.867359. Epub 2013 Dec 16. PMID 24329122